CLINICAL TRIAL: NCT01573806
Title: Phase 1-2 Study of the Pharmacology of Exenatide in Pediatric Sepsis
Brief Title: Pharmacology of Exenatide in Pediatric Sepsis
Acronym: PEPS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jerry Zimmerman, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEPS-SCH-001
Record Dates: First submitted 2012-03-28; First posted 2012-04-10 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Septic Shock; Inflammation; Glucose Homeostasis; Organ Dysfunction; Health-related Quality of Life
Keywords: sepsis; septic shock; children; incretins; exenatide; pharmacokinetics; pharmacodynamics; glucose homeostasis; inflammation; cytokines; health-related quality of life; functional status
MeSH Terms: conditions — Shock, Septic; Inflammation; Sepsis | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Active Comparator): Subjects dosed with exenatide in Phase 2
  Interventions: Drug: Exenatide
- Exenatide vehicle (Placebo Comparator): Subjects dosed with exenatide vehicle in Phase 2
  Interventions: Drug: Exenatide vehicle

INTERVENTIONS:
Drug: Exenatide — Exenatide, dosed subcutaneously every 12 hours for 4 doses
  Arms: Exenatide
Drug: Exenatide vehicle — Exenatide vehicle, dosed subcutaneously every 12 hours for 4 doses
  Arms: Exenatide vehicle

SUMMARY:
Pharmacology of Exenatide in Pediatric Sepsis, PEPS is a phase 1-2 research study that will examine drug safety, drug metabolism, drug action and preliminary drug clinical effects of four does of exenatide injected every 12 hours to children with shock from infection (septic shock). The investigators hypothesize that exenatide can be safely dosed to children with sepsis to achieve blood levels of drug similar to that achieved in teenagers with type 2 diabetes. The investigators further hypothesize that injection of exenatide to children with septic shock will normalize blood glucose levels and decrease levels of inflammation proteins in the blood during the early course of sepsis.

DETAILED DESCRIPTION:
Pharmacology of Exenatide in Pediatric Sepsis, PEPS is a phase 1-2 investigation that will examine safety, pharmacokinetics, pharmacodynamics, and preliminary clinical efficacy of 4 subcutaneous doses of exenatide administered every 12 hours to children with newly diagnosed septic shock. The investigators' long term goal is to explore the potential benefit of exenatide on: early immunomodulation and glucose homeostasis, organ dysfunction, and clinically meaningful outcomes associated with pediatric sepsis. The current study objectives are to conduct a "3+3" dose escalation study, and then examine a "best exenatide allometric dose" to generate safety, pharmacokinetic, pharmacodynamic, and initial efficacy data in a larger cohort. In Phase 1 (three allometric doses; three age strata)the investigators will identify an exenatide dosing regimen that mimics area under the exenatide concentration curve for exenatide dosing among adolescents with type 2 diabetes with minimal or no adverse events. A total of 18 subjects are expected to be enrolled in Phase 1. In Phase 2 the investigators will utilize this "best exenatide allometric dose" to further clarify exenatide safety (adverse event occurence: e.g. nausea, abdominal pain, delayed gastric emptying, hypoglycemia, pancreatitis, renal dysfunction), pharmacokinetics, pharmacodynamics (glucose homeostasis; inflammatory cytokine serum concentrations), and effect on clinical outcomes (AUC of Saturation Index, AUC Vasoactive-Inotropic Score, AUC RIFLE Criteria, Pediatric Logistic Organ Dysfunction Score; changes in health-related quality of life and functional status). In Phase 2, 30 subjects in each age strata in the ratio of 4:1, exenatide: vehicle, are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age 44 weeks estimated gestational age to 18 years AND
* Admitted to the PICU for the sepsis event AND
* Vascular catheter capable of providing serial blood samples in place AND
* Diagnosis of septic shock = sepsis with cardiovascular organ dysfunction AND
* Parents speak English or Spanish

Exclusion Criteria:

* Greater than 12 hours from admission to PICU to enrollment OR
* Chronic or acute dialytic therapy, history of renal impairment or renal transplantation OR
* History of pancreatitis OR
* History of hypersensitivity to Byetta OR
* History of severe gastrointestinal disease or gastroparesis OR
* History of diabetes mellitus, type I or type II OR
* History of insulin, sulfonyl urea drugs, or coumarin use OR
* History of hypoglycemia OR
* History of active pregnancy (effect of exenatide on the fetus is unknown) OR
* Inability to collect serial blood samples OR
* Previously enrolled in the PEPS study OR
* Lack of commitment to aggressive sepsis therapy OR
* Expectation to succumb from the sepsis event OR
* Patient is a foster child and/or ward of the state OR
* Sepsis event associated with a PICU-acquired nosocomial infection OR
* Patient is enrolled in another interventional investigation that might obscure the potential effects of exenatide dosing.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Exenatide associated adverse event occurence | From PICU admission to PICU discharge, an average interval of 7.5 days
  Potential adverse events associated with exenatide: nausea, abdominal pain, hypoglycemia, delayed gastric emptying, pancreatitis, renal dysfunction, reactions at injection site. Adverse event occurence will be tabulated while the subject remains in the PICU.
Exenatide pharmacokinetics: Area under the exenatide concentration curve for 4 subcutaneous exenatide injections administered every 12 hours. | 48 hours following the first exenatide dose
  Delineation of the pharmacokinetics of subcutaneously dosed exenatide among children with de novo septic shock.

SECONDARY OUTCOMES:
Exenatide pharmacodynamics: Effect of exenatide on glucose homeostasis | 60 hours following first exenatide dose
  Delineation of exenatide pharmacodynamics among children with de novo septic shock: AUC of all serum glucose values or results of continuous glucose monitoring obtained during the 60 hours following the first dose of exenatide (or drug vehicle).
Exenatide pharmacodynamics: Effect of exenatide on serum inflammatory cytokine concentrations. | 60 hours following first exenatide dose
  Delineation of exenatide pharmacodynamics among children with de novo septic shock: AUC of serial serum inflammatory cytokine concentrations.
Exenatide clinical efficacy: Effect of exenatide on intensity and duration of organ dysfunctions. | From PICU admission to PICU discharge, an average interval of 7.5 days
  AUC of daily Pediatric Logistic Organ Dysfunction (PELOD) scores while the subject remains in the PICU
Exenatide clinical efficacy: Effect of exenatide on intensity and duration of hemodynamic instability. | From onset to discontinuation of vasoactive-inotropic support, an average interval of 4 days
  AUC of daily Vasoactive-Inotropic Scores while the subject remains on vasoactive-inotropic support.
Exenatide clinical efficacy: Effect of exenatide on intensity and duration of pulmonary failure. | From onset to discontinuation of mechanical ventilator support, an average interval of 4.5 days
  AUC of daily Saturation Indices ([FiO2*MAP]/SpO2)
Exenatide clinical efficacy: Effect of exenatide on intensity and duration of renal failure | From PICU admission to PICU discharge, an average interval of 7.5 days
  AUC of daily RIFLE criteria
Exenatide clinical efficacy: Effect of exenatide on magnitude of sepsis-associated change in functional status. | 2 measurements: baseline and PICU discharge, the latter occuring on average at 7.5 days
  Determination per parent report of declination from baseline to PICU discharge of, Pediatric Overall Performance Category Score and Functional Status Score
Exenatide clinical efficacy: Effect of exenatide on magnitude of sepsis-associated change in health-related quality of life | 2 measurements: baseline and PICU discharge, the latter occuring on average at 7.5 days
  Determination per parent report of declination from baseline to PICU discharge of, Pediatric Quality of Life Inventory, Generic Core Scales, 4.0 (PedsQL)

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Background] Ivy SP, Siu LL, Garrett-Mayer E, Rubinstein L. Approaches to phase 1 clinical trial design focused on safety, efficiency, and selected patient populations: a report from the clinical trial design task force of the national cancer institute investigational drug steering committee. Clin Cancer Res. 2010 Mar 15;16(6):1726-36. doi: 10.1158/1078-0432.CCR-09-1961. Epub 2010 Mar 9. PMID 20215542
- [Background] Mecott GA, Herndon DN, Kulp GA, Brooks NC, Al-Mousawi AM, Kraft R, Rivero HG, Williams FN, Branski LK, Jeschke MG. The use of exenatide in severely burned pediatric patients. Crit Care. 2010;14(4):R153. doi: 10.1186/cc9222. Epub 2010 Aug 11. PMID 20701787
- [Background] Malloy J, Capparelli E, Gottschalk M, Guan X, Kothare P, Fineman M. Pharmacology and tolerability of a single dose of exenatide in adolescent patients with type 2 diabetes mellitus being treated with metformin: a randomized, placebo-controlled, single-blind, dose-escalation, crossover study. Clin Ther. 2009 Apr;31(4):806-15. doi: 10.1016/j.clinthera.2009.04.005. PMID 19446153
- [Background] Deane AM, Chapman MJ, Fraser RJ, Summers MJ, Zaknic AV, Storey JP, Jones KL, Rayner CK, Horowitz M. Effects of exogenous glucagon-like peptide-1 on gastric emptying and glucose absorption in the critically ill: relationship to glycemia. Crit Care Med. 2010 May;38(5):1261-9. doi: 10.1097/CCM.0b013e3181d9d87a. PMID 20228679